CLINICAL TRIAL: NCT03490175
Title: Genetic Variants and Non-genetic Variables Associated With Postoperative Nausea and Vomiting (PONV)
Brief Title: Genetic Variants and Non-genetic Variables and Postoperative Nausea and Vomiting
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 041/09b PONV
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Anesthesia; Analgesia; Surgical Procedure, Operative
Keywords: genetic association study; postoperative nausea and vomiting; patient reported outcome; antiemetics
MeSH Terms: conditions — Agnosia; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (plasma and cells) or mucosal swab
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All patients: Patients undergoing general anesthesia for elective surgery

SUMMARY:
Prospective observational study to analyse the association of non-genetic variables as well as genetic variants of candidate genes with the incidence of postoperative nausea and vomiting (PONV).

DETAILED DESCRIPTION:
Background

Surgery and anesthesia are related to unwanted adverse events, side effects and postoperative discomfort. Postoperative nausea and vomiting are frequent and the question arises which patient is at specific risk for these sequelae. Some predisposing factors for PONV are well described, e.g. female sex, non-smoking status and postoperative opioids. Some drugs used for anesthesia as well as surgery related variables might induce PONV.

In this prospective association study patient related variables, surgical and anesthesia related variables as well as genetic variants of several candidate genes will be investigated in a well-described patient cohort presenting for scheduled surgery.

Objective

The aim of this study is to investigate a possible association of non-genetic variables and genetic variants with PONV.

Methods

Prospective association study performed in patients recovering form elective surgery and anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Written informed consent
* Elective surgery

Exclusion Criteria

* No written informed consent
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 2778 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Association study: genetic and non-genetic variables associated with No PONV, Intermediate PONV and Severe PONV | perioperative period up to 48 hours after surgery
  PONV composite outcome measured by episodes of vomiting and nausea + need for antiemetic treatment + results of a patient reported outcome questionnaire. Patients with no PONV are compared to those with intermediate and severe PONV. Bariatric patients will not be included in this analysis.

SECONDARY OUTCOMES:
Sex specific association analysis: Severity of PONV associated with genetic and non-genetic variables in males and females | perioperative period up to 48 hours after surgery
  PONV composite outcome measured by episodes of vomiting and nausea + need for antiemetic treatment + results of a patient reported outcome. questionnaire. Patients with no PONV are compared to those with intermediate and severe PONV
Association study in patients undergoing bariatric surgery: genetic and non-genetic variables associated with No PONV, Intermediate PONV and Severe PONV | perioperative period up to 48 hours after surgery
  PONV composite outcome measured by episodes of vomiting and nausea + need for antiemetic treatment + results of a patient reported outcome questionnaire. Patients with no PONV are compared to those with intermediate and severe PONV

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Stamer, Prof. MD, Study Chair — Department of Anaestheisology and Pain Medicine, Inselspital, University of Bern; Ulrike M Stamer, MD, Principal Investigator — Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern, Bern, Switzerland

REFERENCES:
- [Derived] Stamer UM, Schmutz M, Wen T, Banz V, Lippuner C, Zhang L, Steffens M, Stuber F. A serotonin transporter polymorphism is associated with postoperative nausea and vomiting: An observational study in two different patient cohorts. Eur J Anaesthesiol. 2019 Aug;36(8):566-574. doi: 10.1097/EJA.0000000000001014. PMID 31274544